CLINICAL TRIAL: NCT05727332
Title: Vascular Adaptations to Single-Sprint Training
Acronym: VASST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Principal Investigator, Matthew Jessee, Assistant Professor, University of Mississippi, Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U54GM115428 (NIH)
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular System
Keywords: Vascular; Cardiorespiratory Fitness

STUDY DESIGN:
Intervention Model Description: Intervention group and negative control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will perform a single maximal effort sprint on a cycle ergometer for twenty seconds 3 days/week for 4 weeks.
  Interventions: Behavioral: Single-Sprint Training
- Time-Matched Control (No Intervention): The control group will be asked to maintain pre-intervention habits/behavior over 4 weeks.

INTERVENTIONS:
Behavioral: Single-Sprint Training — A single maximal effort sprint on a cycle ergometer for twenty seconds 3 days/week for 4 weeks
  Arms: Intervention

SUMMARY:
The long-term objective of this research line is to identify and implement an effective and feasible intervention capable of preventing and/or reducing the burden of cardiometabolic and obesity-related diseases that affect Mississippians and others. The pursuit of this long-term objective will begin with achieving the specific aims proposed in this pilot project, which are to determine the effect of single sprint training for improving (1) systemic macro-vascular function, (2) local and systemic micro-vascular function, and (3) cardiorespiratory fitness. These aims will be achieved using a randomized controlled trial whereby 40 males and females will be randomized into an intervention group (n=20) or time-matched negative control group (n=20). The intervention group will perform a single maximal effort sprint on a cycle ergometer for twenty seconds 3 days/week for 4 weeks and the control group will be asked to maintain pre-intervention habits/behavior over 4 weeks. All outcome measures are non-invasive, and will be assessed pre-, mid-, and post-intervention, with the exception of cardiorespiratory fitness, which will be measured pre- and post-. To achieve aim 1, brachial artery flow-mediated dilation via ultrasonography and systolic and diastolic blood pressure via automated oscillometry will be measured on the arm. To achieve aim 2, post-occlusive reactive hyperemia via near-infrared spectroscopy and reactive hyperemia via ultrasound will be measured in the arm and leg, respectively. To achieve aim 3, pulmonary gas exchange will be measured during a graded exercise test on a cycle ergometer. All outcomes will be compared across time between conditions and sex with a three-way Bayesian Repeated Measures ANOVA using pre-values as covariates and an uninformed prior. 95% credible intervals will also be calculated to power future investigations using this intervention. If the intervention is found effective, future studies will be conducted to determine the efficacy of the intervention in larger groups and more clinical populations, and to determine the mechanisms mediating the adaptations. If ineffective, the knowledge gained will be used to develop future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Untrained (no regular exercise engagement for the previous 6 months)
* Healthy enough to begin exercise (assessed via Physical Activity Readiness Questionnaire)

Exclusion Criteria:

* Illness/injury preventing cycling exercise
* Prescribed medication to control heart rate
* Prescribed medication to control blood pressure
* Use of nicotine within the previous 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline systemic macrovascular function at 2 weeks and 4 weeks | week 0, week 2, and week 4
  Systemic macrovascular changes will be quantified by measuring 1) brachial artery flow-mediated dilation via vascular ultrasound, and 2) resting brachial blood pressure via a standard automated blood pressure cuff.
Change from baseline local and systemic microvascular function at 2 weeks and 4 weeks | week 0, week 2, and week 4
  Systemic changes in microvascular endothelial function will be quantified by using the post-occlusive reactive hyperemia technique in the arm. Local microvascular function will be measured using the passive leg movement technique for reactive hyperemia and post-occlusive reactive hyperemia in the leg.

SECONDARY OUTCOMES:
Change from baseline maximal oxygen consumption at 2 weeks and 4 weeks | week 0, week 2, and week 4
  To assess changes in cardiorespiratory fitness, pulmonary gas exchange data will be collected during a maximal graded exercise test on a cycle ergometer. VO2max and ventilation thresholds will be reported in accordance with current guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual data outside of the investigators responsible for conducting the study. If data are requested, they will only be shared after being de-identified, unless otherwise required by law.